CLINICAL TRIAL: NCT05016804
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Systemic Sclerosis
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell IV Infusion for Systemic Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-10-ATG-12-04
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Systemic Sclerosis
Keywords: Systemic Sclerosis; Scleroderma; stem cell treatment
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Systemic Sclerosis

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Systemic Sclerosis. Patients with Systemic Sclerosis will receive a single intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease requiring chemotherapeutic drugs such as methotrexate, an autologous T Cell vaccine will be utilized created from the patient's own T cells obtained by apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Sclerosis
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: skin score | Four year follow-up
  It will be completed for each follow up point.
Efficacy: Forced vital capacity (FVC) | Four year follow-up
  It will be completed for each follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Center for Investigation in Tissue Engineering and Cellular Therapy, Buenos Aires, Argentina

REFERENCES:
- [Background] Kaldas M, Khanna PP, Furst DE, Clements PJ, Kee Wong W, Seibold JR, Postlethwaite AE, Khanna D; investigators of the human recombinant relaxin and oral bovine collagen clinical trials. Sensitivity to change of the modified Rodnan skin score in diffuse systemic sclerosis--assessment of individual body sites in two large randomized controlled trials. Rheumatology (Oxford). 2009 Sep;48(9):1143-6. doi: 10.1093/rheumatology/kep202. Epub 2009 Jul 14. PMID 19605370
- [Background] Granel B, Daumas A, Jouve E, Harle JR, Nguyen PS, Chabannon C, Colavolpe N, Reynier JC, Truillet R, Mallet S, Baiada A, Casanova D, Giraudo L, Arnaud L, Veran J, Sabatier F, Magalon G. Safety, tolerability and potential efficacy of injection of autologous adipose-derived stromal vascular fraction in the fingers of patients with systemic sclerosis: an open-label phase I trial. Ann Rheum Dis. 2015 Dec;74(12):2175-82. doi: 10.1136/annrheumdis-2014-205681. Epub 2014 Aug 11. PMID 25114060
- [Background] Del Papa N, Di Luca G, Andracco R, Zaccara E, Maglione W, Pignataro F, Minniti A, Vitali C. Regional grafting of autologous adipose tissue is effective in inducing prompt healing of indolent digital ulcers in patients with systemic sclerosis: results of a monocentric randomized controlled study. Arthritis Res Ther. 2019 Jan 7;21(1):7. doi: 10.1186/s13075-018-1792-8. PMID 30616671